CLINICAL TRIAL: NCT06669247
Title: A First-in-Human (FIH) Phase 1/2 Study to Assess Safety, Tolerability, and Preliminary Anti-Tumor Activity of REGN7945, an Anti-CD38 x Anti-CD28 Costimulatory Bispecific Monoclonal Antibody, in Combination With Linvoseltamab, an Anti-BCMA x Anti-CD3 Bispecific Monoclonal Antibody, in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Assess the Safety and Anti-Tumor Activity of REGN7945 in Combination With Linvoseltamab in Adult Participants With Relapsed/Refractory Multiple Myeloma
Acronym: COSTIMM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R7945-ONC-22110; 2024-513126-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: R/RMM
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase 1: non-randomized dose escalation Phase 2: randomized dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- REGN7945+Linvoseltamab (Experimental): Phase 1 Phase 2
  Interventions: Drug: REGN7945+Linvoseltamab
- Linvoseltamab (Experimental): Phase 2
  Interventions: Drug: Linvoseltamab; Drug: REGN7945+Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Administered per protocol
  Other Names: REGN5458
  Arms: Linvoseltamab
Drug: REGN7945+Linvoseltamab — Administered per protocol

SUMMARY:
This study is researching an experimental drug called REGN7945 in combination with another experimental drug called linvoseltamab, (also known as REGN5458) (each individually called a "study drug" or "study drugs" when combined).

This study is the first time REGN7945 will be tested in humans. Linvoseltamab has previously been studied by itself (without other cancer drugs) in participants who had advanced multiple myeloma that returned and needed to be treated again after several other therapies had failed.

The aim of the study is to see how safe, tolerable, and effective REGN7945 is when given in combination with linvoseltamab, compared with linvoseltamab alone.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug(s)
* How many people treated with REGN7945 and linvoseltamab compared to linvoseltamab alone have improvement of their multiple myeloma and by how much
* How long people benefit from receiving REGN7945 in combination with linvoseltamab compared with linvoseltamab alone
* How much study drug(s) is in the blood at different times
* Whether the body makes antibodies against the study drugs(s) (which could make the study drug(s) less effective or could lead to side effects)
* If there is any change in pain and cancer-related symptoms, how well people are able to function, and their quality of life when taking the study drug(s)

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤1 as described in the protocol
2. Received at least 3 lines of therapy including exposure to at least 1 anti-CD38 antibody, 1 immunomodulatory imide drug (IMiD), and 1 proteasome inhibitor (PI) and have demonstrated disease progression on or after the last therapy, as defined in the protocol. Prior treatment with other BCMA directed immunotherapies, including BCMA CAR-T cells and BCMA antibody-drug conjugates (Phase 1 and 2), and with BCMA x CD3 bispecific antibodies (Phase 1 only), is allowed
3. Participants must have the measurable disease for response assessment as described in the protocol
4. Adequate hematologic, hepatic, and renal function as described in the protocol

Key Exclusion Criteria:

1. Diagnosis of plasma cell leukemia, primary systemic light-chain amyloidosis (including myeloma associated amyloidosis), Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
2. Treatment with any systemic anti-cancer therapy within 5 half-lives or within 28 days before first administration of study drug, whichever is shorter
3. History of allogeneic stem cell transplantation within 6 months, or autologous stem cell transplantation within 12 weeks of the start of study treatment
4. Treatment with systemic corticosteroid treatment with more than 10 mg per day of prednisone or steroid equivalent within 72 hours of start of study drug
5. Participants who have known central nervous system (CNS) involvement with MM or known or suspected progressive multifocal leukoencephalopathy (PML), history of a neurocognitive condition or CNS disorder, or history of seizure within 12 months prior to study enrollment
6. Live or live attenuated vaccination within 28 days before first study drug administration with a vector that has replicative potential
7. Has received a COVID-19 vaccination within 1 week of planned start of study medication as described in the protocol
8. Myelodysplastic syndrome or another malignancy in the past 3 years, except for nonmelanoma skin cancer, in situ carcinoma, thyroid cancer, or low-risk early stage prostate adenocarcinoma, as described in the protocol
9. Significant cardiovascular disease as described in the protocol
10. Uncontrolled infection with HIV, Hep B or Hep C infection, or other uncontrolled infection, such as CMV, as described in the protocol
11. Known hypersensitivity to both allopurinol and rasburicase

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2033-11-11 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) from the first dose of REGN7945 in combination with linvoseltamab | Up to 21 days
  Phase 1
Incidence of treatment emergent adverse events (TEAEs) during the treatment period with REGN7945 in combination with linvoseltamab | Up to 5 years
  Phase 1
Severity of TEAEs during the treatment period with REGN7945 in combination with linvoseltamab | Up to 5 years
  Phase 1
Very Good Partial Response (VGPR) or better as determined by the investigator using the International Myeloma Working Group (IMWG) response criteria in patients receiving combination therapy | Within 12 weeks of starting cycle 1
  Phase 2
VGPR or better as determined by the investigator using the IMWG response criteria in patients receiving linvoseltamab monotherapy | Within 12 weeks of starting cycle 1
  Phase 2
Partial Response (PR) or better as determined by the investigator using the IMWG response criteria in patients receiving combination therapy | Within 12 weeks of starting cycle 1
  Phase 2
PR or better as determined by the investigator using the IMWG response criteria in patients receiving linvoseltamab monotherapy | Within 12 weeks of starting cycle 1
  Phase 2

SECONDARY OUTCOMES:
Incidence of TEAEs | Up to 5 years
  Phase 1 and Phase 2
Severity of TEAEs | Up to 5 years
  Phase 1 and Phase 2
Concentrations of REGN7945 in the serum | Up to 5 years
  Phase 1 and Phase 2
Concentrations of linvoseltamab in the serum | Up to 5 years
  Phase 1 and Phase 2
Incidence of anti-drug antibodies (ADA) to REGN7945 | Up to 5 years
  Phase 1 and Phase 2
Titer of ADA to REGN7945 | Up to 5 years
  Phase 1 and Phase 2
Incidence of ADA to linvoseltamab | Up to 5 years
  Phase 1 and Phase 2
Titer of ADA to linvoseltamab | Up to 5 years
  Phase 1 and Phase 2
Change in European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30) Global Health Status / Quality of Life (GHS/QoL) | Up to 5 years
  Phase 1 and Phase 2 The EORTC QLQ-C30 is a 30-item validated questionnaire developed to measure patient-reported quality of life using one global health status/quality of life (GHS/QoL) scale, 5 functioning scales (physical, role, emotional, cognitive, and social) ranging from from 1 = "very poor" to 5 = "excellent" and 9 symptom scales/items (fatigue, nausea/vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) among patients with cancer, ranging from 1 = "not at all" to 9 = "very much" higher scores indicate higher symptom burden.
Change in EORTC QLQ-C30 Physical Functioning (PF) | Up to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-C30 Role Functioning (RF) | Up to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-C30 pain | Up to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-C30 fatigue | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-C30 GHS/QoL | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-C30 PF | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-C30 RF | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-C30 pain | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-C30 fatigue | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-C30 GHS/QoL | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-C30 PF | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-C30 RF | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-C30 pain | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-C30 fatigue | Up to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-Multiple Myeloma Module (MY20) Disease Symptoms (DS) | Up to 5 years
  Phase 1 and Phase 2 The EORTC QLQ-MY20 is a self -administered instrument to assess QoL in persons with Multiple Myeloma (MM). This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item). A high score represents a high level of symptoms or problems.
Change in EORTC QLQ-MY20 Treatment Side Effects (TSE) | Up to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-MY20 Body Image (BI) | UP to 5 years
  Phase 1 and Phase 2
Change in EORTC QLQ-MY20 Future Perspective (FP) | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-MY20 DS | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-MY20 TSE | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-MY20 BI | Up to 5 years
  Phase 1 and Phase 2
Time to definitive deterioration in EORTC QLQ-MY20 FP | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-MY20 DS | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-MY20 TSE | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-MY20 BI | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EORTC QLQ-MY20 FP | Up to 5 years
  Phase 1 and Phase 2
Change in EuroQoL-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) Visual Analogue Score (VAS) (EQ-5D-5L VAS) | Up to 5 years
  Phase 1 and Phase 2 The EQ-5D-5L is a generic questionnaire that measures Health-Related Quality of Life (HRQoL) across 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) across 5 levels (no problems, slight problems, some problems, severe problems and extreme problems) and a visual analogue scale (VAS).
Time to definitive deterioration in EQ-5D-5L VAS | Up to 5 years
  Phase 1 and Phase 2
Time to first improvement in EQ-5D-5L VAS | Up to 5 days
  Phase 1 and Phase 2
Patient-reported overall impact of treatment toxicity measured by Functional Assessment of Cancer Therapy (FACIT)-Item GP5 | Up to 5 years
  Phase 1 and Phase 2 FACIT-Item GP5 will be used to assess the patient-reported impact of treatment toxicity that uses a single item "I am bothered by side effects of treatment" on a 5-point scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much).
Objective Response Rate (ORR) as measured by IMWG criteria as determined by the investigator | Up to 5 years
  Phase 1
Complete response (CR) rate as measured by IMWG criteria as determined by the investigator | Up to 5 years
  Phase 1
Duration of response (DOR) by IMWG criteria as determined by the investigator | Up to 5 years
  Phase 1
Progression Free Survival (PFS) as measured by IMWG criteria as determined by the investigator | Up to 5 years
  Phase 1
Achievement of Minimal Residual Disease (MRD) negative status (at 10^5) in participants in CR or better | Up to 5 years
  Phase 1
Overall survival (OS) | Up to 5 years
  Phase 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (7):
- Australia (5):
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Alfred Hospital, Melbourne, Victoria
- United Kingdom (2):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/